CLINICAL TRIAL: NCT02491814
Title: The Effect of Commercially-available Dairy and Non-dairy Alternatives When Consumed With a High Glycemic Cereal on Subjective Appetite Ratings and Post-meal Glycemia in Healthy Young Adults
Brief Title: The Effect of Dairy and Non-dairy Alternatives on Satiety and Post-meal Glycemia in Healthy Young Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DFC_31012
Record Dates: First submitted 2015-05-27; First posted 2015-07-08 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes; Obesity
Keywords: Dairy; Breakfast cereal; Postprandial Glycemia; Satiety; Food Intake; Milk; Yogurt; Soy; Almond
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Milk; Soy Milk; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1% M.F. Milk and Breakfast Cereal (Experimental): Breakfast meal: 250 ml 1% M.F. Milk, 54 g Cheerios breakfast cereal, 100 mL water
  Interventions: Other: 1% M.F. Milk; Other: Breakfast cereal
- Yogurt Beverage and Breakfast Cereal (Experimental): Breakfast meal: 250 ml Yogurt Beverage, 54 g Cheerios breakfast cereal, 100 mL water
  Interventions: Other: Yogurt Beverage; Other: Breakfast cereal
- Soy Beverage and Breakfast Cereal (Experimental): Breakfast meal: 250 ml Soy Beverage, 54 g Cheerios breakfast cereal, 100 mL water
  Interventions: Other: Soy Beverage; Other: Breakfast cereal
- Almond Beverage and Breakfast Cereal (Experimental): Breakfast meal: 250 ml Almond Beverage, 54 g Cheerios breakfast cereal, 100 mL water
  Interventions: Other: Almond Beverage; Other: Breakfast cereal
- Water (control) and Breakfast Cereal (Experimental): Breakfast meal: 250 ml Water, 54 g Cheerios breakfast cereal, 100 mL water
  Interventions: Other: Water; Other: Breakfast cereal

INTERVENTIONS:
Other: 1% M.F. Milk
  Other Names: 1% cow's milk; Neilsen Canada
  Arms: 1% M.F. Milk and Breakfast Cereal
Other: Yogurt Beverage
  Other Names: Yop (Vanilla), General Mills
  Arms: Yogurt Beverage and Breakfast Cereal
Other: Soy Beverage
  Other Names: Soy Milk; Silk Organic Original
  Arms: Soy Beverage and Breakfast Cereal
Other: Almond Beverage
  Other Names: Almond Milk; Silk Original
  Arms: Almond Beverage and Breakfast Cereal
Other: Water
  Other Names: Calorie-free control
  Arms: Water (control) and Breakfast Cereal
Other: Breakfast cereal
  Other Names: Cheerios, General Mills

SUMMARY:
This study investigates the effects of commercially-available dairy (1% cow's milk and yogurt beverage) and non-dairy alternatives (almond and soy beverages) on satiety and post-meal blood glucose. Each participant will receive every treatment in this crossover design study.

DETAILED DESCRIPTION:
Regular consumption of dairy is associated with better body composition and lower incidences of type 2 diabetes and obesity. This may be due to dairy's ability to increase satiety and decrease post-prandial glycemia. However, most clinical studies have only investigated isolated dairy proteins (whey and casein) and the effects of whole dairy products remains unclear. Additionally, as non-dairy alternatives are becoming more popular there is interest to see if they can elicit similar benefits as dairy. Therefore, this study will test the effects of commercially-available dairy and non-dairy beverages when consumed with cereal at breakfast time.

Thirty healthy young males and females (20-30 years, BMI 20.0-24.9 kg/m2) will be recruited for the randomized, unblinded, crossover study. Participants will fast overnight, and at baseline will consume 250 mL of 1% milk, soy beverage, almond beverage, yogurt beverage, or water with 54 g of Cheerios cereal. At 0 (baseline), 15, 30, 45, 60, 75, 90, 120 minutes (pre-meal period) 140, and 170 minutes (post-meal period) blood will be collected for glucose analysis and subjective appetite ratings completed. Insulin will be analyzed every 30 minutes and for the last two timepoints. Between 120-140 minutes, an ad libitum lunch will be provided to assess food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy BMI (20.0 - 24.9 kg/m2)
* Females with regular monthly menstrual cycles

Exclusion Criteria:

* Diabetes
* Fasting blood glucose higher than 5.8 mmol/L
* Pregnancy
* Medications
* Smoking
* Lactose intolerance or allergies to milk, soy, or almonds
* Elite athletes
* Those trying to lose or gain weight
* Breakfast skippers and those on an energy-restricted diet
* Score equal to or higher than 11 on Eating Habits Questionnaire

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 0-170 minutes
  Blood glucose (mmol/L) is measured using finger prick capillary blood samples
Subjective Appetite | 0-170 minutes
  Subjective appetite ratings are obtained from four 100 mm visual analogue scale (VAS) questions assessing "Desire to Eat", "Hunger", "Fullness" and "Prospective Food Consumption". The average of all four VAS is calculated to obtain the average appetite score for statistical analysis

SECONDARY OUTCOMES:
Insulin | 0-170 minutes
  Blood insulin (μU/mL) is measured using finger prick capillary blood samples
Food Intake | 120-140 minutes
  Food at an ad libitum pizza lunch will be weighed to determine food intake based on nutrition information provided by the pizza manufacturer

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, Ph.D., Principal Investigator — Department of Nutritional Sciences, University of Toronto
Locations (1):
- Department of Nutritional Sciences, FitzGerald Building, Toronto, Ontario, Canada